CLINICAL TRIAL: NCT04555785
Title: Enhancement of the Haemostatic Effect of Platelets in the Presence of High Normal Concentrations of Von Willebrand Factor
Acronym: Will-Plate
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-02106
Record Dates: First submitted 2020-08-25; First posted 2020-09-21 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — von Willebrand Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet transfusion with Wilate ® (Experimental)
  Interventions: Drug: Wilate
- Platelet transfusion with Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Wilate — Wilate ® will be given with platelets in cases of severe bleeding. Wilate ® is a 1:1 balanced mixture of von Willebrand Factor (2'000 IU) and Coagulation factor VIII (2'000 IU) and as such has anti-haemorrhagic potential. It is extracted from plasma, freeze-dried and virus-inactivated.
  Arms: Platelet transfusion with Wilate ®
Other: Placebo — Empty placebo will be given with platelets in cases of severe bleeding.
  Arms: Platelet transfusion with Placebo

SUMMARY:
Assessment of high-normal dosage of Wilate ® compared to placebo administered in combination with platelets to assess reduction of amount of blood loss, need of transfusion products and outcome (length of stay, mortality) in patients with bleeding in comparison.

DETAILED DESCRIPTION:
Von Willebrand Factor (vWF) is a key protein mediating platelet adhesion on the surface of damaged endothelia, initiating platelet-platelet aggregation and supporting platelet activation. It plays also an important role in protecting FVIII from early activation and clearance . The product's included coagulation factor VIII acts in in the activated form like the regular factor VIIIa. It takes part in the coagulation amplification by activating factor X to Xa together with factor IVa. Activation of factor X results in generating thrombin out of prothrombin. Wilate® is approved in Switzerland for prophylaxis and treatment of bleeding in patients suffering from von Willebrand disease and Haemophilia A.

VWF is produced by the endothelial cells as a heterogeneous mixture of low and high molecular weight units. VWF is a ligand for receptors on the platelet surface and endothelial cells (GP1b-V-IX, αIIbβ3, αvβ3) mediating adhesion of platelets to each other or to the endothelium. Initial platelet adhesion is a crucial step in haemostatic functioning. Loss of platelets, vWF or blocking of these integrins due to the wide use of platelet aggregation inhibitors can cause bleeding. In case of severe blood loss, these conditions often result in mass transfusion.

There is suggestive evidence from an in-vitro flow chamber model and from treatment of patients with severe vWF deficiency that increasing the concentration of vWF onto normal or high normal levels can enhance platelet adhesion independent from platelet count. This might translate into a better haemostatic effect of administered platelet concentrates in the bleeding patient and less need for transfusion of blood products (platelet concentrates), especially in clinical conditions with a high probability of low platelet count and low vWF activities (e.g., heart surgery with extracorporeal circulation, ECMO).

To the best of our knowledge, no trial exists that investigated the effect of platelet transfusion in combination with the administration of balanced vWF in severe blood loss. The investigators hypothesize that simultaneous transfusion of platelets and balanced (1:1 vWF and FVIII) vWF compared to placebo reduces the overall need of transfusion of blood products.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to intensive care unit
* Patients needing platelet transfusion during or after surgery with or without prior treatment with single or dual antiplatelet agents (ASS, Prasugrel, Clopidogrel, Ticagrelor)
* Consent by the patient or a family member in addition to the consent of an independent ICU physician

Exclusion Criteria:

* Patients receiving Factor VIII concentrate before inclusion of the study (Haemate ®)
* Women who are pregnant or breastfeeding
* Participation in another study with an investigational drug within the 30 days preceding and during the present study
* Overt Disseminated Intravascular Coagulation (DIC)
* Heparin-induced Thrombocytopenia (HIT)
* Thrombotic Thrombocytopenic Purpura (TTP) or Haemolytic uremic Syndrome (HUS)
* Idiopathic thrombocytopenic purpura (ITP)
* Sepsis
* Patients with known inherited thrombocytopathies
* Patients with known von Willebrand disease or Haemophilia A
* Patients with known hemato-oncological diseases
* Previous enrolment into the current study
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of blood products | 48 hours
  Number of blood products (fresh frozen plasma (FFP), red blood cells (RBC)) according to groups.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Siegemund, Prof. Dr. MD, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ledergerber K, Hollinger A, Zimmermann S, Todorov A, Trutmann M, Gallachi L, Gschwandtner LA, Ryser LA, Gebhard CE, Bolliger D, Buser A, Tsakiris DA, Siegemund M. Impact of Additional Administration of von Willebrand Factor Concentrates to Thrombocyte Transfusion in Perioperative Bleeding in Cardiac Surgery. Transfus Med Hemother. 2023 Jul 11;51(1):22-31. doi: 10.1159/000530810. eCollection 2024 Feb. PMID 38314243
- [Derived] Herrmann G, Blum A, Bolliger D, Achermann R, Estermann A, Gebhard CE, Henn A, Huber J, Singh J, Todorov A, Zehnder T, Zellweger N, Buser A, Tsakiris DA, Hollinger A, Siegemund M. Enhancement of the haemostatic effect of platelets in the presence of high normal concentrations of von Willebrand factor for critically ill patients needing platelet transfusion-a protocol for the will-plate randomised controlled trial. Trials. 2023 Jan 20;24(1):47. doi: 10.1186/s13063-022-06876-8. PMID 36670471